CLINICAL TRIAL: NCT00953108
Title: Impact of Quetiapine Prolong and Escitalopram on the Hypothalamic-pituitary-adrenocortical (HPA)-Axis Activity in Depressed Patients
Brief Title: Quetiapine Prolong, Escitalopram and Hypothalamic-pituitary-adrenocortical (HPA) Axis Activity in Depressed Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Cornelius.Schuele, MD, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QUE/09
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Quetiapine Fumarate; Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- quetiapine (Experimental)
  Interventions: Drug: quetiapine
- escitalopram (Active Comparator)
  Interventions: Drug: escitalopram

INTERVENTIONS:
Drug: quetiapine — 300 mg per day
  Arms: quetiapine
Drug: escitalopram — escitalopram 10 mg per day
  Arms: escitalopram

SUMMARY:
In former studies of the investigators research group the investigators could also demonstrate acute inhibitory effects of the antidepressant mirtazapine on ACTH and cortisol release in normal controls (Schüle et al. 2002), most likely mediated via antagonism at central 5-HT2- and H1-receptors. In contrast to mirtazapine, serotonin or norepinephrine reuptake inhibiting antidepressants acutely stimulate ACTH and cortisol secretion (Schüle 2007). The investigators also performed a study in depressed patients who were treated either with mirtazapine or with reboxetine using serial dexamethasone/CRH tests (week 0, 1, and 5) as a parameter for HPA axis activity. Mirtazapine, but not the norepinephrine reuptake inhibitor reboxetine was able to significantly reduce HPA axis activity already within one week (Schüle et al. 2006). Mirtazapine is known to have an earlier onset of antidepressant action than do SSRIs such as sertraline (Behnke et al. 2003) or antidepressants with dual mechanism of action such as venlafaxine (Benkert et al. 2006), possibly due to its rapid inhibition of HPA axis activity in unipolar depressed patients.

Since mirtazapine and quetiapine have similar effects on the HPA system in healthy male volunteers (i.e. inhibition of ACTH and cortisol secretion), a rapid attenuation of HPA axis activity is also expected during quetiapine XR treatment in depressed patients.

Therefore, in the present study the investigators goal is to investigate whether quetiapine fumarate XR at a dosage of 300 mg per day has an impact on HPA axis activity in unipolar depressed patients, as measured by serial dexamethasone/CRH tests (week 0, 1, and 5) and salivary cortisol profiles and whether putative effects of quetiapine XR on the HPA system are related to its antidepressant efficacy.

ELIGIBILITY:
Inclusion criteria:

For inclusion in the study patients must fulfil all of the following criteria:

1. Inpatients (the admission to hospital occurs independently from study participation)
2. Provision of written informed consent
3. A diagnosis of major depression by Diagnostic and Statistical Manual of Mental Disorders- Fourth Edition (DSM-IV) (unipolar depression: 296.2, 296.3)
4. Female and male patients aged 18 to 65 years
5. Female patients of childbearing potential must have a negative serum human chorionic gonadotropin (hCG) pregnancy test at enrolment and e willing to use a reliable method of birth control (i.e. barrier method, oral contraceptive, implant, dermal contraception, long-term injectable contraceptive, intrauterine device, or tubal litigation) during the study.
6. Able to understand and comply with the requirements of the study as judged by the investigator.
7. A sum score of at least 18 on the 21-item version of the Hamilton Depression Rating Scale (21-HAMD)

Exclusion criteria:

Any of the following is regarded as a criterion for exclusion from the study:

1. Pregnancy or lactation
2. Any DSM-IV Axis I disorder not defined in the inclusion criteria
3. Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
4. Known intolerance or lack of response to quetiapine fumarate and/or escitalopram, as judged by the investigator
5. Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrolment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir
6. Use of any of the following cytochrome P450 3A4 inducers in the 14 days preceding enrolment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids
7. Use of monoamine oxidase inhibitors (MAOIs) or other serotonergic drugs (e.g. triptans) in the 14 days preceding enrolment
8. Use of oral anticoagulants in the 14 days preceding enrolment
9. History of bleeding disorders.
10. Use of drugs which are mainly metabolized by cytochrome P450 2D6 having a low therapeutic index (e.g. flecainide, propafenone, metoprolol) in the 14 days preceding enrolment
11. Administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomisation
12. Substance or alcohol dependence at enrolment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by DSM-IV criteria
13. Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM-IV criteria within 4 weeks prior to enrolment
14. Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
15. Unstable or inadequately treated medical illness (e.g. congestive heart failure, angina pectoris, hypertension) as judged by the investigator
16. Involvement in the planning and conduct of the study
17. Previous enrolment or randomisation of treatment in the present study.
18. Participation in another drug trial within 4 weeks prior enrolment into this study or longer in accordance with local requirements
19. A patient with Diabetes Mellitus (DM) fulfilling one of the following criteria:

    * Unstable DM defined as enrolment glycosylated hemoglobin (HbA1c) >8.5%.
    * Admitted to hospital for treatment of DM or DM related illness in past 12 weeks.
    * Not under physician care for DM
    * Physician responsible for patient's DM care has not indicated that patient's DM is controlled.
    * Physician responsible for patient's DM care has not approved patient's participation in the study
    * Has not been on the same dose of oral hypoglycaemic drug(s) and/or diet for the 4 weeks prior to randomisation. For thiazolidinediones (glitazones) this period should not be less than 8 Weeks.
    * Taking insulin whose daily dose on one occasion in the past 4 weeks has been more than 10% above or below their mean dose in the preceding 4 weeks Note: If a diabetic patient meets one of these criteria, the patient is to be excluded even if the treating physician believes that the patient is stable and can participate in the study.
20. An absolute neutrophil count (ANC) of 1.5 x 109 per liter
21. Abnormal laboratory parameters of clinical relevance before enrolment
22. Abnormal blood pressure, abnormal electrocardiogram, and/or abnormal electroencephalogram with clinical relevance before enrolment
23. Psychotropic drugs within 3 days before and throughout the study with the exception of zopiclon (up to 7.5 mg per day) in case of sleep difficulties and lorazepam (up to 2 mg per day) in case of inner tension and anxiety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
serial dexamethasone/CRH tests | week 0, 1, and 5

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, Ludwig-Maximilian-University, Munich, Bavaria, Germany

REFERENCES:
- [Derived] Sarubin N, Nothdurfter C, Schmotz C, Wimmer AM, Trummer J, Lieb M, Uhr M, Baghai TC, Wetter TC, Buhner M, Rupprecht R, Schule C. Impact on cortisol and antidepressant efficacy of quetiapine and escitalopram in depression. Psychoneuroendocrinology. 2014 Jan;39:141-151. doi: 10.1016/j.psyneuen.2013.10.008. Epub 2013 Oct 23. PMID 24275013